CLINICAL TRIAL: NCT01882933
Title: GASTRICHIP : D2 Resection and HIPEC (Hyperthermic Intraperitoneal Chemoperfusion) in Locally Advanced Gastric Carcinoma. A Randomized and Multicentric Phase III Study.
Brief Title: D2 Resection and HIPEC (Hyperthermic Intraperitoneal Chemoperfusion) in Locally Advanced Gastric Carcinoma
Acronym: GASTRICHIP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012.761
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric adenocarcinoma; HIPEC; Oxaliplatin; Signet ring cell
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curative Gastrectomy + HIPEC (Experimental): Curative gastrectomy with D1-D2 lymph node dissection + HIPEC with oxaliplatin
  Interventions: Drug: HIPEC (Hyperthermic Intraperitoneal Chemoperfusion) with oxaliplatin; Procedure: Curative gastrectomy
- Curative Gastrectomy (Other): Curative gastrectomy with D1-D2 lymph node dissection
  Interventions: Procedure: Curative gastrectomy

INTERVENTIONS:
Drug: HIPEC (Hyperthermic Intraperitoneal Chemoperfusion) with oxaliplatin — After the D2 resection is complete HIPEC can start. A roller pump forces the chemotherapy solution (oxaliplatin 250 mg/m² with 2 Liters of G5%/m²) into the abdomen through the inflow catheter and pulls it out through the drains. A heat exchanger keeps the intraperitoneal fluid at 42°-43°C.
  Arms: Curative Gastrectomy + HIPEC
Procedure: Curative gastrectomy — All the patients will undergo a D1-D2 gastrectomy carried out according to Japanese guidelines and to the European recommendations for the preservation of spleen and pancreas

SUMMARY:
A prospective, opened, multicentric, randomised, phase III trial with two arms:

* Arm A: curative gastrectomy with D1-D2 lymph node dissection + HIPEC with oxaliplatin
* Arm B: curative gastrectomy with D1-D2 lymph node dissection

Main objective: Compare overall 5-year survival rates in patients surgically treated for advanced gastric adenocarcinoma (T3, T4 and/or N+ and/or with positive peritoneal cytology), treated either with curative gastrectomy and adjuvant HIPEC, or with curative gastrectomy alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 75 years old
* White blood cells > 3,500/mm3, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3
* Good renal functions, serum creatinine values being < 1.5 mg/dl and creatinine clearance > 60 ml/min
* Performance Status ≤1, Karnofsky Index ≥ 70%
* Serum bilirubin ≤ 2 mg/dl
* Having given written informed consent prior to any procedure related to the study.
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research
* Not under any administrative or legal supervision
* Histologically evidenced resectable T3 or T4 gastric adenocarcinoma for which a curative gastrectomy is scheduled, with invasion into the serosa AND/OR lymph node metastasis (determined from data obtained by endoscopic ultrasound and chest, abdomen and pelvis CT scan) AND/OR positive peritoneal cytology (sampled during the preoperative laparoscopy).

AND/OR

* Perforated gastric adenocarcinoma AND/OR
* Siewert III adenocarcinoma of the cardia for which a gastrectomy by exclusive abdominal laparotomy is scheduled
* Females of childbearing age potential and male subjects with partners of childbearing potential using efficient contraceptive measures (as judged by the investigator).Subjects randomised in the arm with HIPEC should be informed and accept that these requirements should also extend to :

  * 4 months after the treatment with Oxaliplatin for female subjects,
  * 6 months after the treatment with Oxaliplatin for male subjects.

Exclusion Criteria:

* Prior malignant tumors with detectable signs of recurrence
* Gastric stump adenocarcinoma
* Presence of comorbidities, notably serious chronic diseases or organ failure General conditions
* Any subject in exclusion period of a previous study according to applicable regulations
* Pregnancy or breastfeeding
* Females of childbearing age potential or male subjects with partners of childbearing potential not using medically accepted contraceptive measures, as judged by the investigator Interfering substance
* Contraindication to any drug contained in the chemotherapy regimen Specific to the study
* Life threatening toxicity before surgery
* Distant metastases (liver, lung. ovaries, etc)
* Tumoral infiltration of the head or body of the pancreas
* Patients presenting an adenocarcinoma of the cardia Siewert I or II
* Existence of macroscopic peritoneal implants
* Patients with clinically significant ascites (> 500 cc) even if cytology is negative for cancer cells, in the absence of other non-malignant causes of ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  From the date of surgery to the date of death or to the end of follow-up

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
  From the date of surgery to the date of recurrence or to the end of follow-up
Recurrence-free survival | 3 years
  From the date of surgery to the date of recurrence or to the end of follow-up
Locoregional-free survival | 5 years
  From the date of surgery to the date of locoregional recurrence or to the end of follow-up
Treatment-related morbidity | During the 60th postoperative days
  Common Terminology Criteria for Adverse Events v4.0
Treatment-related mortality | During the 60th postoperative days
Score QLQ-C30 | 3 months (M3), 6 months (M6) and 12 months (M12) after surgery +/- HIPEC procedure.
  Quality of life is assessed with EORTC questionnaire QLQ-C30
Score QLQ-STO 22 | 3 months (M3), 6 months (M6) and 12 months (M12) after surgery +/- HIPEC procedure.
  Quality of life is assessed with EORTC questionnaire QLQ-STO 22

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GLEHEN, MD, Principal Investigator — Service de Chirurgie Générale Digestive et Endocrinienne, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon
Locations (33):
- France (27):
  - Département de Chirurgie Digestive, CHU d'Amiens, Amiens
  - Service de Chirurgie Digestive Oncologique, CLCC Paul Papin, Angers
  - Département de Chirurgie Digestive - CHU d'Angers, Angers
  - Service de Chirurgie Digestive, Hôpital Jean Minjoz, CHU Besançon, Besançon
  - Service de Chirurgie Viscérale, CLCC François Baclesse, Caen
  - Service de Chirurgie Viscérale, CHU Estaing, Clermont-Ferrand
  - Service de Chirurgie Digestive, Hôpital du Bocage, Dijon
  - Service de Chirurgie Digestive et de l'Urgence, Hôpital Michallon, Grenoble
  - Service de Chirurgie Digestive et Générale, Hôpital Huriez, Lille
  - Service de Chirurgie Digestive, CLCC Léon Bérard, Lyon
  - Service d'Oncologie Digestive, Hôpital de la Timone, Marseille
  - Service de Chirurgie Digestive, CRLC Val d'Aurelle, Montpellier
  - Service de Chirurgie Digestive, CLCC René Gauducheau, Nantes
  - Service de Chirurgie Digestive, Hôpital Archet II, Nice
  - Service de Chirurgie Digestive, Institut Curie, Paris
  - Service de Chirurgie Viscérale et Oncologique, Hôpital Saint-Louis, Paris
  - Service de Chirurgie Générale et Digestive, Hôpital Saint-Antoine, APHP, Paris
  - Service de Chirurgie Digestive, Hôpital Lariboisière, Paris
  - Service de Chirurgie Générale Digestive et Endocrinienne, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Service de Chirurgie Viscérale, CHU de Poitiers, Poitiers
  - Service de Chirurgie Générale et Viscérale, CHU de Reims - Hôpital Robert Debré, Reims
  - Service de Chirurgie Digestive et de Physiologie Digestive, Hôpital Ch. Nicolle, Rouen
  - Service de Chirurgie Digestive, Hôpital Nord, Saint-Etienne
  - Service de Chirurgie Viscérale et Digestive, Hôpital de Hautepierre, Strasbourg
  - Service de Chirurgie Générale et Digestive, Hôpital Purpan, Toulouse
  - Service de Chirurgie Digestive Oncologique, CLCC Alexis Vautrin, Vandœuvre-lès-Nancy
  - Département de Chirurgie Digestive et Hépatobiliaire, Institut Gustave Roussy, Villejuif
- Spain (6):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares
  - Hospital Sant Joan Despí Moises Broggi, Barcelona
  - Md Anderson Cancer Center, Madrid
  - Fundación Jiménez Díaz Hospital, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid

REFERENCES:
- [Derived] Glehen O, Passot G, Villeneuve L, Vaudoyer D, Bin-Dorel S, Boschetti G, Piaton E, Garofalo A. GASTRICHIP: D2 resection and hyperthermic intraperitoneal chemotherapy in locally advanced gastric carcinoma: a randomized and multicenter phase III study. BMC Cancer. 2014 Mar 14;14:183. doi: 10.1186/1471-2407-14-183. PMID 24628950